CLINICAL TRIAL: NCT07198607
Title: The Role of Pistacia Lentiscus Oil as a Preventive Tool for Chronic Rhinosinusitis Recurrence in Long-Term Therapy: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Pistacia Lentiscus Oil Nasal Drops for Preventing Recurrence of Chronic Rhinosinusitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Collaborators: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental Medicine, Liaquat University of Medical & Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IAR20221123
Record Dates: First submitted 2025-09-15; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Chronic Rhinosinusitis Without Nasal Polyps; Chronic Rhinosinusitis (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: Participants were randomized in a 1:1 ratio to receive either isotonic saline wash plus Pistacia lentiscus oil nasal drops or isotonic saline wash plus placebo drops.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind trial in which participants, care providers, investigators, and outcome assessors were unaware of group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Pistacia lentiscus Oil Nasal Drops (Experimental): Participants will receive isotonic saline nasal wash plus Pistacia lentiscus oil nasal drops. Dosage: 5 drops per nostril twice daily for 30 days, followed by maintenance therapy of 5 drops per nostril twice daily for 15 days each month over the subsequent 11 months.
  Interventions: Other: Pistacia lentiscus Oil Nasal Drops (Bactorinol®)
- Placebo Comparator: Placebo Nasal Drops (Placebo Comparator): Participants will receive isotonic saline nasal wash plus placebo nasal drops, matched in appearance and administration schedule. Dosage: 5 drops per nostril twice daily for 30 days, followed by maintenance therapy of 5 drops per nostril twice daily for 15 days each month over the subsequent 11 months.
  Interventions: Other: Placebo Nasal Drops (matched to Bactorinol®)

INTERVENTIONS:
Other: Pistacia lentiscus Oil Nasal Drops (Bactorinol®) — Bactorinol® nasal drops (medical device containing ultra-fractioned and winterized Pistacia lentiscus oil). Participants will receive isotonic saline nasal wash plus 5 drops per nostril twice daily for 30 days, followed by 5 drops per nostril twice daily for 15 days per month for the subsequent 11 months.
  Other Names: Winterized Pistacia lentiscus oil; Bactorinol®
  Arms: Experimental: Pistacia lentiscus Oil Nasal Drops
Other: Placebo Nasal Drops (matched to Bactorinol®) — Placebo nasal drops identical in appearance and administration to Bactorinol®. Participants will receive isotonic saline nasal wash plus placebo drops, 5 drops per nostril twice daily for 30 days, followed by 5 drops per nostril twice daily for 15 days per month for the subsequent 11 months.
  Other Names: Saline-based placebo drops
  Arms: Placebo Comparator: Placebo Nasal Drops

SUMMARY:
This randomized, double-blind, placebo-controlled clinical trial evaluated the safety and efficacy of nasal drops containing Pistacia lentiscus oil in preventing recurrence of chronic rhinosinusitis. Adult patients with chronic rhinosinusitis were randomized 1:1 to receive either isotonic saline wash plus Pistacia lentiscus oil drops or isotonic saline wash plus placebo, for a total treatment duration of 12 months. The primary outcome was change in Sino-Nasal Outcome Test-22 (SNOT-22) scores, while secondary outcomes included ciliary motility, nasal secretion, biofilm presence, cytological changes, adverse events, and safety/tolerability.

DETAILED DESCRIPTION:
Chronic rhinosinusitis (CRS) is a common and recurrent condition associated with significant morbidity and impaired quality of life. Standard treatment approaches often provide only partial or temporary relief, and recurrence rates remain high. Pistacia lentiscus oil has demonstrated anti-inflammatory and mucosal protective properties, supporting its potential role as a preventive intervention in CRS management.

This monocenter, non-profit, randomized, placebo-controlled trial was designed to evaluate the long-term preventive effect of Pistacia lentiscus oil nasal drops on CRS recurrence. One hundred patients aged ≥18 years with diagnosed CRS were randomized in a 1:1 ratio to either the intervention group (isotonic saline wash plus Pistacia lentiscus oil drops, 5 drops per nostril twice daily for 30 days, followed by maintenance treatment for 15 days per month over 11 months) or the placebo group (isotonic saline wash plus placebo drops on the same schedule).

The primary endpoint was the change in disease-specific quality of life, measured by the Sino-Nasal Outcome Test-22 (SNOT-22) from baseline to 12 months. Secondary endpoints included assessments of ciliary motility, nasal secretion, presence of biofilm, supranuclear striae, bacterial cells, variations in inflammatory cellularity (neutrophils, eosinophils, mast cells), safety, and tolerability. The study received ethical approval from the Italian Academy of Rhinology (Ref: IAR20221123).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Clinical diagnosis of chronic rhinosinusitis
* Nasal polypoid score ≤1
* ≥4 episodes of recurrence per year
* SNOT-22 score ≥10 Willingness and ability to provide written informed consent

Exclusion Criteria:

* Nasal polypoid score >2
* <4 episodes of recurrence per year
* SNOT-22 score <10
* Known immune disorders
* Neoplastic disorders
* Neurological disorders
* Psychiatric disorders
* Inability to undergo treatment
* Refusal or inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Sino-Nasal Outcome Test-22 (SNOT-22) score | Baseline, 1 month, and 1 year
  The SNOT-22 questionnaire measures disease-specific quality of life in chronic rhinosinusitis patients. Scores range from 0 (no symptoms) to 110 (worst symptoms).

SECONDARY OUTCOMES:
Ciliary motility | Baseline, 1 month, and 1 year
  Assessment of ciliary beat frequency and duration using phase contrast optical microscopy; considered normal if beating lasts >10 minutes.
Presence of Nasal Secretion | Baseline, 1 month, and 1 year
  Presence or absence of nasal secretion, assessed by anterior rhinoscopy.
Characteristics of Nasal Secretion | Baseline, 1 month, and 1 year
  Nasal secretion characteristics (clear, mucopurulent, or purulent) will be graded by anterior rhinoscopy using standardized clinical evaluation.
Presence of biofilm | Baseline, 1 month, and 1 year
  Cytological evaluation of mucosal samples stained for biofilm, identified by cyan-colored areas.
Presence of supranuclear striae | Baseline, 1 month, and 1 year
  Microscopic evaluation of nasal mucosa samples for supranuclear striae.
Presence of bacterial cells | Baseline, 1 month, and 1 year
  Cytological evaluation of mucosal samples for bacterial cells.
Cellularity variation | Baseline, 1 month, and 1 year
  Quantitative cytology of neutrophils, eosinophils, and mast cells from nasal mucosa samples.
Number of Participants With Treatment-Related Adverse Events | Throughout study period (up to1 year)
  Safety will be assessed by recording all adverse events (local and systemic) related to nasal drop use, as evaluated by the investigator.
Local Tolerability of Nasal Drops | Baseline, 1 month, and 1 year
  Local tolerability will be assessed by anterior rhinoscopy for signs of nasal irritation (redness, swelling, mucosal damage) and patient-reported nasal discomfort using a Visual Analogue Scale (0-10).

CONTACTS AND LOCATIONS:
Locations (1):
- Ent Clinic ASST Settelaghi, University of Insubriae, Varese, Italy

IPD SHARING:
Plan to Share IPD: No